CLINICAL TRIAL: NCT03110016
Title: Feasibility, Usability, User Satisfaction, and Preliminary Efficacy of a Smartphone Intervention for Subthreshold Depression
Brief Title: Smartphone Intervention for Subthreshold Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kibi International University (Other)
Responsible Party: Principal Investigator, Kazuki Hirao, PhD, OT, Assistant Professor, Kibi International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16-55
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Subthreshold Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone Application (Experimental): SPSRS is a smartphone application system designed to improve self-confidence in individuals with subthreshold depression. The application presents a motion picture that displays words every 5 s for improving self-confidence of the user.
  Interventions: Device: Smartphone Application

INTERVENTIONS:
Device: Smartphone Application — The participants use SPSRS to watch the motion picture for at least 10 min a day for 5 weeks.

SUMMARY:
The study aimed to examine the feasibility, usability, user satisfaction, safety, and preliminary efficacy of a smartphone application intervention for young adults with subthreshold depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-24 years
* Has a Center for Epidemiologic Studies Depression Scale score of ≥16
* Owns a smartphone with the iOS® operating system

Exclusion Criteria:

* Lifetime history of major depressive disorder
* Lifetime history of bipolar disorder
* Currently receiving treatment for a mental health problem from a mental health professional
* Experience of a major depressive episode in the 2 weeks prior to the study, as ascertained using the Mini-International Neuropsychiatric Interview

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility, as measured by adherence to the smartphone application intervention. | 5 weeks after initiating the intervention
  Adherence is calculated as the number of minutes in a week for which the participant uses the SPSRS application divided by the recommended weekly duration (70 min).

SECONDARY OUTCOMES:
Usability and user satisfaction | 5 weeks after initiating the intervention
  USE Questionnaire
Number of participants with treatment-related adverse events as assessed by Mini-International Neuropsychiatric Interview. | baseline and 1, 2, 3, 4, and 5 weeks after initiating the intervention
  Mini-International Neuropsychiatric Interview
Depressive symptoms | baseline and 5 weeks after initiating the intervention
  Center for Epidemiologic Studies Depression Scale score
Inflammatory biomarker | baseline and 5 weeks after initiating the intervention
  Level of salivary interleukin-6
General self-efficacy | baseline and 5 weeks after initiating the intervention
  General Self-Efficacy Scale score
Social anxiety | baseline and 5 weeks after initiating the intervention
  Liebowitz Social Anxiety Scale score
Mental health | baseline and 5 weeks after initiating the intervention
  12-item General Health Questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Hirao, PhD, Principal Investigator — Kibi International University
Locations (1):
- Kibi International University, Takahashi, Okayama-ken, Japan